CLINICAL TRIAL: NCT04547608
Title: The Impact of the Timing of Rocuronium After Induction With Propofol on Temporal Summation of Pain in Gynecologic Laparoscopic Surgery-prospective and Controlled Study.
Brief Title: Timing of Rocuronium After Induction With Propofol on Temporal Summation of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WonkwangUH7
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Gynecological Disorder
Keywords: Pain, Propofol, Rocuronium, Temporal summation.
MeSH Terms: conditions — Genital Diseases, Female; Pain

STUDY DESIGN:
Intervention Model Description: One hundred patients, between 18-60 years of age were randomly assigned to one of the two groups; group PRi received immediate injection of rocuronium after propofol administration, and group PRd received rocuronium injection when bispectral index score became below 60 after propofol administration
Who Masked: Outcomes Assessor
Masking Description: Attending anesthesiologist knew which anesthetic agents were used. However Outcomes assessor didn't know which anesthetic agents were used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group PRi (Other): received immediate injection of rocuronium after propofol administration,
  Interventions: Other: The difference of the timing of rocuronium administration after propofol injection
- group PRd (Other): rocuronium injection when bispectral index score became below 60 after propofol administration
  Interventions: Other: The difference of the timing of rocuronium administration after propofol injection

INTERVENTIONS:
Other: The difference of the timing of rocuronium administration after propofol injection — The difference of the timing was rocuronium was administered immediately after propofol injection or when BIS score became below 60 after propofol administration.

SUMMARY:
Temporal summation of pain, which is defined as the perception of increasingly greater pain evoked by repetitive painful stimuli, is highly variable between individuals. This study aimed to determine the impact of the timing of rocuronium after induction with propofol on temporal summation of pain in gynecologic laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective gynecologic laparoscopic surgery
* American Society of Anesthesiologists' physical status class) I-II

Exclusion Criteria:

* Menopause (to exclude the hormonal effect on pain)
* Patients who had muscular, cardiovascular, hepatic or kidney disorders and patients with a history of medication who would affect muscle relaxants were excluded from this study.
* Patients with difficult venous access on forearm, a known allergy to propofol or rocuronium, chronic pain, pregnancy, and those who had received analgesics or sedatives within the previous 24 hours, were excluded from the study.

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — to exclude the hormonal effect on pain
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
the grade of rocuronium induced withdrawal movement. | during anesthesia induction
  withdrawal movements were graded by the investigator according to the following scale:
  1. - no pain (no response);
  2. - mild pain (movement at wrist only);
  3. - moderate pain (movement involving the arm only with elbow or shoulder);
  4. - severe pain (generalized response or movement in more than one extremity

SECONDARY OUTCOMES:
visual analog scale (VAS) for injection pain | during anesthesia induction
  check VAS for pain after propofol administration. visual analog scale with 100 mm for pain after surgery. 0 = no pain, 100 = the worst pain
VAS for pain | at 1 hour, 24 hours and 48 hours
  check VAS with 100 mm for pain after surgery. 0 = no pain, 100 = the worst pain
Patient controlled analgesia (PCA) Opioid consumption | at 24 and 48 hours
  check the volume of PCA Opioid consumption (ml) (PCA) pump containing fentanyl (800 ug), ketorolac (150 mg), and ramosetron (0.6 mg) in a total volume of 150 mL of saline was set to deliver a basal infusion of 2 mL/h and bolus doses of 0.5 mL, with a 15-min lockout period for postoperative analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D,Ph.D, Study Director — Department of anesthesiology and pain medicine
Locations (1):
- WonwangUH, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng JC, Erpelding N, Kucyi A, DeSouza DD, Davis KD. Individual Differences in Temporal Summation of Pain Reflect Pronociceptive and Antinociceptive Brain Structure and Function. J Neurosci. 2015 Jul 1;35(26):9689-700. doi: 10.1523/JNEUROSCI.5039-14.2015. PMID 26134651
- [Background] Ayoglu H, Altunkaya H, Ozer Y, Yapakci O, Cukdar G, Ozkocak I. Does dexmedetomidine reduce the injection pain due to propofol and rocuronium? Eur J Anaesthesiol. 2007 Jun;24(6):541-5. doi: 10.1017/S0265021506002250. Epub 2007 Jan 23. PMID 17241503
- [Background] Hwang SM, Cho SH, Lim SY, et al. The efficacy of BIS monitoring for the preventing of withdrawal movement on the intravenous injection of rocuronium. Korean J Anesthesiol 2005;49:293-7.
- [Background] Lim BG, Lee IO, Kim YS, Won YJ, Kim H, Kong MH. The utility of bispectral index monitoring for prevention of rocuronium-induced withdrawal movement in children: A randomized controlled trial. Medicine (Baltimore). 2017 Jan;96(2):e5871. doi: 10.1097/MD.0000000000005871. PMID 28079825